CLINICAL TRIAL: NCT04972214
Title: The Influence of Infant Feeding Type on Preterm Infant's Intestinal Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Hye-Rim Kim, professor, CHA University
Other Study IDs: 2021-03-062-004
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Microbial Colonization
Keywords: intestinal microbiota; very preterm infant; breast milk; preterm formula
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples are directly collected from the diaper every 14 days for 28 days. Samples are frozen and stored at -80'C for later analysis. DNA will be extracted from the fecal samples, and different bacterial genus and species will be quantified by real-time polymerase chain reaction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Very Preterm Infants: preterm infants were born at gestational age of less than 32 weeks

SUMMARY:
This study aims to examine the factors associated with preterm infant's intestinal microbiota depending on feeding type (breast milk or preterm formula)

DETAILED DESCRIPTION:
The gut microbiome has been increasingly found to affect human health. Feeding plays an important role in determining the composition and diversity of the neonatal gut microbiome. Preterm infants are at a high risk of gut microbiota disruption and dysbiosis because of physiological immaturity and environmental factors. In preterm infants, breast milk has been associated with improved growth and cognitive development and a reduced risk of necrotizing enterocolitis and late onset sepsis.

The objective of study is to determine the impact of feeding type on gut microbiome of very preterm infants admitted in a neonatal intensive care unit (NICU). Meconium and the additional 2 fecal samples will be collected from preterm infants. Fecal samples will be collected every 14 days, during 28 days, from diapers into sterile tubes. DNA will be extracted from fecal samples and different bacterial genus and species will be analyzed.

The type of infant feeding (breast milk or preterm formula) is recorded daily to classify the type of infant feeding received during the 14 days prior to each fecal sample collection.

ELIGIBILITY:
Inclusion Criteria:

- Very preterm infants (< 32 weeks gestational age) admitted in the NICU of CHA Bundang Medical Center within the first 24 hours after birth

Exclusion Criteria:

* Parents refuse to participate/sign informed consent
* Major congenital anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Very preterm infants born before 32 gestational weeks and admitted to the NICU of CHA Bundang Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
intestinal microbiome composition according to the type of feeding | within 24 hours after birth
  comparison of intestinal microbiome with 16s RNA gene specific sequencing in stool
intestinal microbiome composition according to the type of feeding | 2 weeks after birth
  comparison of intestinal microbiome with 16s RNA gene specific sequencing
intestinal microbiome composition according to the type of feeding | 4 weeks after birth
  comparison of intestinal microbiome with 16s RNA gene specific sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Hye-Rim Kim, MD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No